CLINICAL TRIAL: NCT02479165
Title: Pain Management After Cardiac Surgery - Opioids or NSAID? A Randomized Prospective Study
Brief Title: Pain Management After Cardiac Surgery - Opioids or NSAID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Martin Agge Nørgaard, MD, DMsc, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The NSAID trial
Record Dates: First submitted 2015-03-31; First posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Postoperative Pain; Renal Insufficiency; Myocardial Infarction
MeSH Terms: conditions — Pain, Postoperative; Renal Insufficiency; Myocardial Infarction | interventions — Ibuprofen; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Opioid group (Active Comparator): If randomized to the opiod group, the patient was given the following regimen for 1 week, upon return from the intensive care unit, after surgery.
  Tbl. Oxycodone (slow-release) 10mg, Twice daily for 1 week Tbl. Paracetamol 1000mg, Four times daily for 1 week Tbl.oxycodone 5mg Max 4 times daily, as needed, until discharge. Inj, oxycodone 2.5 mg, Max 4 times daily, as needed, until discharge Tbl. Magnesia 1g, Twice daily, for 1 week Sol. Sodiumpicosulfate 7.5mg/ml 10 drops daily, for 1 week
  Interventions: Drug: Oxycodone
- Ibuprofene group (Active Comparator): If randomized to the ibuprofen group, the patient was given the following regimen for 1 week, upon return from the intensive care unit, after surgery.
  Tbl. Ibuprofen (slow-release) 800mg, Twice daily, for 1 week Tbl. Paracetamol 1000mg, Four times daily, for 1 week Tbl.oxycodone 5mg Max 4 times daily, as needed. Until discharge. Inj, oxycodone 2.5 mg Max 4 times daily, as needed. Until discharge. Tbl. Lanzoprazole 40 mg, Once daily, for 1 week Tbl. Magnesia 1g, Twice daily, for 1 week Sol. Sodiumpicosulfate 7.5mg/ml, 10 drops daily, for 1 week
  Interventions: Drug: Ibuprofene

INTERVENTIONS:
Drug: Ibuprofene — The Ibuprofene group is given an ibuprofen based analgesic regimen, to be compared with the standard opiod based regimen.
  Other Names: Ipren; Advil; Motrin; Nurofen
  Arms: Ibuprofene group
Drug: Oxycodone — The opioid group is given an oxycodone based analgesic regimen.
  Other Names: Oxycontin
  Arms: Opioid group

SUMMARY:
The aim of this randomized controlled study is to shed light on the analgesic properties and side-effect profile of an opiod-based regimen as opposed to an Ibuprofene based regimen.

DETAILED DESCRIPTION:
Background:

Postoperative pain following median sternotomy can represent a major postoperative problem as it can lead to reduced mobilization and shallow, restricted breathing and insufficient cough, which can lead to pulmonary complications.

However, pain management with opioids has frequent side-effects such as confusion, respiratory depression, sedation, nausea and obstipation/ paralytic ilieus. Non-steroid anti-inflammatory drugs (NSAIDs) can been used as opiod-sparing analgesics following cardiac surgery. However, this remains controversial, as NSAIDs has been linked to an increased risk of myocardial infarction, especially in patients with ischaemic heart disease, renal failure, gastrointestinal bleeding, and possibly impaired sternal healing.

The investigators wanted to investigate the analgesic properties of a opiod-based regimen with that of an ibuprofene-based, through randomization of patients to one of the two arms.

Intervention:

The participants were given analgesics in accordance to their randomization group upon return from the postoperative ICU stay.

The opioid regimen relied on a basic dose of slow-release oxycodone ("Oxycontin", Norpharma, Vedbaek, Denmark, 10mg two times daily) and paracetamol ("Panodil", GlaxoSmithKline, Copenhagen, Denmark, 1g four times daily). For "break-through pain" extra oxycodone was administered as injections or capsules (5mg pr. dose). Furthermore laxatives were co-administered to prevent obstipation.

In the ibuprofene regimen slow-release ibuprofen ("Brufen Retard", Abbott, Copenhagen, Denmark, 800mg two times daily) replaced oxycodone as the basic analgesic. In the ibuprofene regimen lansoprazol ("Lansoprazole", Actavis, Gentofte, Denmark, 30mg once daily) was co-administered to prevent development of gastric ulcers. These regimens were initiated the first postoperative day, when the patient was transferred from the ICU to the ward, and continued until the seventh postoperative day. Some patient

Outcome:

Please refer to the "outcome" chapter

Statistics:

Data are presented as number of patients, medians, and ranges. Patients are compared according to the ibuprofen or the oxycodone group, and statistics were done using "intention-to-treat"-design. Fischer's exact test, Mann-Whitney, and 95% confidence intervals were used as appropriate. Significance was defined as P-values below 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery through median sternotomy
* Written consent
* Age over 18 years

Exclusion Criteria:

* Other forms of sternotomy (i.e. re-sternotomy or partial sternotomy)
* Preoperative creatinine over 110 µmol/L
* Preoperative use of opioids or NSAIDs in analgesic doses (aspirin in antithrombotic doses was accepted)
* Allergy to NSAIDs or opioids, and other contraindications to the used drugs

The postoperative exclusion criteria were:

* Staying more than one night at the intensive care unit
* Unacceptable side effects
* Exclusion at the patients request

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Pain score - Visual Analouge Scale | 5 days
  Visual analouge scale from 0-10, recorded at noon every day. Given as average/minimum/maximum previous 24h by patient. Until discharge, average 5th postoperative day.

SECONDARY OUTCOMES:
Bowel movement, hours until movement | 5 days
  Time is noted of first bowel movement. Registration until discharge, average 5th postoperative day.
Nausea, Hours | 5 days
  At noon, the total hours of nausea over the previous 24h is noted. Registration until discharge, average 5th postoperative day.
Vomiting, events pr. 24 hours | 5 days.
  Number of themes the patient has vomitted is noted. Registration until discharge, average 5th postoperative day.
Hallucination, events pr. 24 hours | 5 days
  At noon, it is recorded wether the patient has experienced hallucinations the previous 24h. Registration until discharge, average 5th postoperative day.
Confusion | 5 days
  At noon, it is recorded wether the patient can name the given time, physical location own social security number. Registration until discharge, average 5th postoperative day.
Opioid antidote | 5 days
  At noon, it is recorded if the patient is given opiod antagonists (such as Naloxone) the previous 24h. Registration until discharge, average 5th postoperative day.
Renal function as serum-creatinine (micromol/l) | 36 months
  Se-creatinine recorded on the morning of postoperative day 1, 2 and 4 and as out-patient at followup.
Myocardial Infarction, no. of cases | 36 months
  Postoperative myocardial infarction according to ESC/ACC/AHA/WHF consensus-report. Registration until discharge, average 5th postoperative day, and as outpatients until followup.
All cause mortality | 36 months
  All cause mortality until followup.
Sternal non-union, no of cases | 36 months
  Sternal non-union from 1 month after surgery until followup.
Gastro-intestinal bleeding, no. of cases | 36 months
  Bleeding verified through gastroscopi or colonoscopi from operation until followup.
Degree of mobilization, Mobilization scale | 5 days
  At noon, the degree of mobilization is noted on an scale from 0 (complete immobilization) - 4 (complete mobilization). Registration until discharge, average 5th postoperative day.

CONTACTS AND LOCATIONS:
Overall Officials: Martin A Norgaard, DMsc, Principal Investigator — Dep. of cardiothoracic surgery, Aalborg university hospital, Denmark